CLINICAL TRIAL: NCT02724319
Title: Implementation of CYP2C19 Genotyping to Guide Antiplatelet Therapy for Patients Undergoing Cardiac Catheterization at UF Health Jacksonville
Brief Title: Implementation of CYP2C19 Genotyping to Guide Antiplatelet Therapy
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201703131; U01HG007269 (NIH); IRB201703131 (Other: Univeristy of Florida)
Record Dates: First submitted 2016-03-08; First posted 2016-03-31 (Estimated); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention; clopidogrel; loss-of-function allele
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — As part of the study, patients will also be asked to provide consent for the collection and storage of a blood sample to be deidentified and stored in the UF College of Pharmacy Center for Pharmacogenomics Bank (IRB 201500133) for future research to examine additional genetic determinants of effectiveness of antiplatelet therapy as well as asked to consent to the sharing of their de-identified research data through database of Genotypes and Phenotypes (dbGaP) .
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Left heart catheterization patients: Patients presenting to the UF Health Jacksonville cardiac catheterization laboratory for left heart catheterization for suspected coronary artery disease and intent to undergo percutaneous coronary intervention will be targeted for enrollment and will be genotyped by SpartanRX
  Interventions: Device: SpartanRX

INTERVENTIONS:
Device: SpartanRX — A buccal swap genetic sample will be collected from eligible patients who provide written informed consent for CYP2C19 testing. Genotyping will be performed by the SpartanRX system as a clinical test at the UF Health Pathology Laboratory in Jacksonville.

SUMMARY:
It is well established that clopidogrel-induced antiplatelet effects is suboptimal in many patients who are thus exposed to an increased risk of adverse cardiovascular events. Studies have shown that genotypes of the cytochrome P450 (CYP) 2C19 enzyme, which is a key determinant of clopidogrel metabolism, contribute to these findings. Prasugrel and ticagrelor are alternative agents whose effectiveness is not dependent on CYP2C19 genotype. A boxed warning on the Food and Drug Administration (FDA)-approved clopidogrel labeling warns of reduced effectiveness in patients with the LOF genotype and recommends alternative therapies in these patients. The availability of an assay recently approved by the FDA, SpartanRX, which provides results within one-hour facilitates performing genetic testing as a clinical test in real-world practice. We therefore propose to 1) examine the feasibility of implementing CYP2C19 genotyping using SpartanRX as standard of care for patients undergoing cardiac catheterization at UF Health Jacksonville providing the opportunity for clinicians to embrace genotype-guided antiplatelet therapy in those who proceed to PCI and 2) determine if CYP2C19 genotype-guided antiplatelet therapy reduces the risk for major adverse cardiovascular outcomes after PCI.

DETAILED DESCRIPTION:
Dual antiplatelet therapy with aspirin and a P2Y12 receptor inhibitor represents the standard of care treatment for the prevention of major adverse cardiovascular events in patients undergoing percutaneous coronary intervention (PCI). Currently, 3 oral P2Y12 receptor inhibitors (clopidogrel, prasugrel, and ticagrelor) are available for clinical use. Clopidogrel remains the most broadly used P2Y12 receptor inhibitor. However, it is well established that clopidogrel-induced antiplatelet effects is suboptimal in many patients who are thus exposed to an increased risk of adverse cardiovascular events. Studies have shown that genotypes of the cytochrome P450 (CYP) 2C19 enzyme, which is a key determinant of clopidogrel metabolism, contribute to these findings. In fact, clopidogrel is a prodrug that requires bioactivation by the CYP2C19 enzyme. Approximately 30-40% of individuals have the loss-of-function (LOF) CYP2C19 genotype and cannot sufficiently convert clopidogrel to its active form, thereby gaining little to no benefit from the drug. Prasugrel and ticagrelor are alternative agents whose effectiveness is not dependent on CYP2C19 genotype. A boxed warning on the Food and Drug Administration (FDA)-approved clopidogrel labeling warns of reduced effectiveness in patients with the LOF genotype and recommends alternative therapies in these patients. Guidelines from the Clinical Pharmacogenetics Implementation Consortium (CPIC) specifically recommend prasugrel or ticagrelor over clopidogrel for patients with a LOF CYP2C19 genotype who undergo PCI. In turn, these recommendations have led to the use in clinical practice of genetic testing of CYP2C19 genotypes as an aid to clinicians in determining therapeutic strategies for patients undergoing PCI. However, the uptake of genetic testing in real-world clinical practice has been limited by the availability of assays able to provide genetic results in a timely fashion. The availability of an assay recently approved by the FDA, SpartanRX, which provides results within one-hour facilitates performing genetic testing as a clinical test in real-world practice. We therefore propose to 1) examine the feasibility of implementing CYP2C19 genotyping using SpartanRX as standard of care for patients undergoing cardiac catheterization at UF Health Jacksonville providing the opportunity for clinicians to embrace genotype-guided antiplatelet therapy in those who proceed to PCI and 2) determine if CYP2C19 genotype-guided antiplatelet therapy reduces the risk for major adverse cardiovascular outcomes after PCI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Undergoing left heart catheterization for signs and symptoms suggestive for CAD

Exclusion Criteria:

* Inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the UF Health Jacksonville cardiac catheterization laboratory for left heart catheterization for suspected coronary artery disease (CAD) and intent to undergo PCI will be targeted for enrollment.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Percent of patients approached who consent to study participation and are genotyped successfully | 48 hours
  Patients undergoing elective procedures will be approached for CYP2C19 genetic testing prior to undergoing left heart catheterization, while patients requiring emergent procedures will be tested prior to hospital discharge.

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | 12 months
  A composite rate of death, myocardial infarction, stroke, stent thrombosis, and ischemia-driven revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Principal Investigator — University of Florida College of Medicine-Jacksonville
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Patients will be asked to also have a single blood sample collected which will be stored for future research, and the option to share data to the public NIH database of Genotypes and Phenotypes (dbGaP). dbGaP was developed to archive and distribute the data and results from studies that have investigated the interaction of genotype and phenotype in Humans.

REFERENCES:
- [Derived] Cavallari LH, Franchi F, Rollini F, Been L, Rivas A, Agarwal M, Smith DM, Newsom K, Gong Y, Elsey AR, Starostik P, Johnson JA, Angiolillo DJ. Clinical implementation of rapid CYP2C19 genotyping to guide antiplatelet therapy after percutaneous coronary intervention. J Transl Med. 2018 Apr 11;16(1):92. doi: 10.1186/s12967-018-1469-8. PMID 29642909